CLINICAL TRIAL: NCT02283788
Title: A Randomized, Double-blind, Placebo-controlled and Open Label Active-controlled, 4-period Crossover Trial to Evaluate the Effect of Eslicarbazepine Acetate on Cardiac Repolarization in Healthy Adult Men and Women
Brief Title: Trial to Evaluate the Effect of Eslicarbazepine Acetate on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-116
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence ABCD (Experimental): A - BIA 2-093 1200 mg once daily × 5 days B - BIA 2-093 2400 mg once daily × 5 days C - Moxifloxacin 400 mg × 1 dose D - placebo once daily × 5 days
  Interventions: Drug: BIA 2-093; Drug: Moxifloxacin; Drug: Placebo
- Treatment Sequence BDAC (Experimental): A - BIA 2-093 1200 mg once daily × 5 days B - BIA 2-093 2400 mg once daily × 5 days C - Moxifloxacin 400 mg × 1 dose D - placebo once daily × 5 days
  Interventions: Drug: BIA 2-093; Drug: Moxifloxacin; Drug: Placebo
- Treatment Sequence CADB (Experimental): A - BIA 2-093 1200 mg once daily × 5 days B - BIA 2-093 2400 mg once daily × 5 days C - Moxifloxacin 400 mg × 1 dose D - placebo once daily × 5 days
  Interventions: Drug: BIA 2-093; Drug: Moxifloxacin; Drug: Placebo
- Treatment Sequence DCBA (Experimental): A - BIA 2-093 1200 mg once daily × 5 days B - BIA 2-093 2400 mg once daily × 5 days C - Moxifloxacin 400 mg × 1 dose D - placebo once daily × 5 days
  Interventions: Drug: BIA 2-093; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate
Drug: Moxifloxacin
  Other Names: avalox
Drug: Placebo
  Other Names: PLC

SUMMARY:
A randomized, double-blind, placebo-controlled and open label active-controlled, 4 period crossover trial to evaluate the effect of eslicarbazepine acetate on cardiac repolarization in healthy adult men and women

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, placebo-controlled and open label active-controlled, 4 period crossover study was to evaluate the effect of therapeutic and supra-therapeutic doses of eslicarbazepine acetate on the placebo corrected time-matched change from baseline using individually corrected QT (QTcI) interval durations in adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male or female 18 to 45 years of age. Women were required to be postmenopausal (more than 12 months since last period); surgically sterile (hysterectomy or tubal ligation at least 6 months prior to enrollment); using an intrauterine device; or double barrier (i.e. diaphragm or spermicide plus male condom) non-hormonal contraceptive therapy for the duration of the trial and were required to have a negative pregnancy test at screening and upon each check-in to the study facility.
* Have a BMI within the range of 18-30 kg/m2.
* Be able to communicate effectively with the study personnel.
* Have no significant disease or abnormal laboratory values as determined by medical history, physical examination or laboratory evaluations, conducted at the screening visit and on each admission to the clinic.
* Have a normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction.
* Be nonsmokers defined as not having smoked in the past 6 months.
* Be adequately informed of the nature and risks of the study and give written informed consent prior to study entry.

Exclusion Criteria:

* Known hypersensitivity or allergy to moxifloxacin, eslicarbazepine acetate or related compounds such as carbamazepine, oxcarbazepine, or licarbazepine.
* Women who were pregnant or breast feeding.
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or placed the subject at increased risk.
* A sustained supine systolic blood pressure > 140 mmHg or <100mm Hg or a diastolic blood pressure > 95 mmHg at screening or baseline.
* A resting ECG heart rate of <50 bpm or >100 bpm.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Phase OneTM, Miramar, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence ABCD: Period 1 - BIA 2-093 1200 mg once daily × 5 days Period 2 - BIA 2-093 2400 mg once daily × 5 days Period 3 - Moxifloxacin 400 mg × 1 dose Period 4 - placebo once daily × 5 days
- Treatment Sequence BDAC: Period 1 - BIA 2-093 2400 mg once daily × 5 days Period 2 - placebo once daily × 5 days Period 3 - BIA 2-093 1200 mg once daily × 5 days Period 4 - Moxifloxacin 400 mg × 1 dose
- Treatment Sequence CADB: Period 1 - Moxifloxacin 400 mg × 1 dose Period 2 - BIA 2-093 1200 mg once daily × 5 days Period 3 - placebo once daily × 5 days Period 4 - BIA 2-093 2400 mg once daily × 5 days
- Treatment Sequence DCBA: Period 1 - placebo once daily × 5 days Period 2 - Moxifloxacin 400 mg × 1 dose Period 3 - BIA 2-093 2400 mg once daily × 5 days Period 4 - BIA 2-093 1200 mg once daily × 5 days
Period: Overall Study
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BDAC | Treatment Sequence CADB | Treatment Sequence DCBA
Started | 17 | 17 | 17 | 16
Completed | 16 | 13 | 12 | 14
Not Completed | 1 | 4 | 5 | 2
Not completed — Adverse Event | 1 | 3 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Sequence ABCD; Treatment Sequence BDAC; Treatment Sequence CADB; Treatment Sequence DCBA: A - BIA 2-093 1200 mg once daily × 5 days B - BIA 2-093 2400 mg once daily × 5 days C - Moxifloxacin 400 mg × 1 dose D - placebo once daily × 5 days
  BIA 2-093
  Moxifloxacin
  Placebo
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BDAC | Treatment Sequence CADB | Treatment Sequence DCBA | Total
Number analyzed (Participants) | 17 | 17 | 17 | 16 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (7.55) | 33.6 (6.41) | 32.6 (7.88) | 35.8 (7.35) | 34.5 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 10 | 9 | 35
  Male | 10 | 8 | 7 | 7 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 4 | 1 | 9
  White | 13 | 16 | 13 | 15 | 57
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: QTcI - QT Interval Individually Corrected for Heart Rate - Day 5
Time Frame: -30 minutes (pre-dose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, and 23.5 hours post-dose
Measure: Mean (Standard Deviation); unit: msec
Groups:
- BIA 2-093 1200 mg; BIA 2-093 2400 mg: ESL, Eslicarbazepine 1200 mg
- Moxifloxacin 400 mg: brand names Avelox, Avalox, and Avelon
- Placebo: Placebo, PLC
Arm/Group | BIA 2-093 1200 mg | BIA 2-093 2400 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 61 | 58 | 61 | 64
msec
  0.5 hr | -8.05 (12.168) | -6.15 (10.891) | -2.77 (10.496) | -4.39 (9.985)
  1 hour | -9.34 (11.399) | -7.34 (11.822) | 3.80 (11.824) | -4.14 (9.515)
  1.5 hours | -8.70 (11.689) | -8.67 (10.525) | 5.30 (11.537) | -4.22 (10.432)
  2 hours | -9.48 (10.692) | -8.31 (10.738) | 6.87 (11.477) | -5.32 (10.189)
  3 hours | -8.04 (11.188) | -8.50 (13.142) | 8.49 (12.875) | -3.24 (11.178)
  4 hours | -7.72 (12.496) | -6.16 (13.563) | 10.13 (11.686) | -2.10 (9.899)
  5 hours | -3.54 (11.282) | -1.71 (12.567) | 7.07 (11.309) | -0.75 (10.090)
  6 hours | -4.59 (11.792) | -2.64 (12.856) | 5.83 (10.927) | -3.10 (10.537)
  8 hours | -2.63 (10.841) | -1.36 (11.281) | 5.80 (12.303) | -1.77 (10.586)
  12 hours | -0.01 (9.347) | 0.03 (13.311) | 5.85 (9.955) | -1.44 (9.150)
  16 hours | -3.72 (10.863) | -4.65 (12.930) | 5.21 (10.900) | -1.41 (12.835)
  23.5 hours | -3.36 (11.514) | -0.06 (12.605) | 2.39 (9.104) | -1.71 (9.513)

2. Secondary Outcome: QTcB - QT Interval Corrected for Heart Rate Using Bazett's Formula
Time Frame: -30 minutes (pre-dose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, and 23.5 hours post-dose
Reporting Status: Not Posted

3. Secondary Outcome: QTcF - QT Interval Corrected Using Fridericia's Formula
Time Frame: -30 minutes (pre-dose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, and 23.5 hours post-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BDAC | Treatment Sequence CADB | Treatment Sequence DCBA
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/17 | 3/17 | 5/17 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Sequence ABCD (N=17) | Treatment Sequence BDAC (N=17) | Treatment Sequence CADB (N=17) | Treatment Sequence DCBA (N=16)
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
dizziness (Nervous system disorders) | 1 | 3 | 5 | 1
Paraesthesia oral (Nervous system disorders) | 0 | 3 | 3 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 3 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 3 | 5 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
VASODILATATION (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other